CLINICAL TRIAL: NCT04628572
Title: Retrospective Analysis to Characterize the Real World Use Patterns, Efficacy and Safety of Ceftazidime-avibactam in the Management of Gram Negative Infections.
Brief Title: Retrospective Analysis of Real World Use of Ceftazidime-avibactam in the Management of Gram Negative Infections
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: X9001260
Record Dates: First submitted 2020-10-07; First posted 2020-11-13 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-02

CONDITIONS: Gram Negative Infections
MeSH Terms: interventions — avibactam, ceftazidime drug combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort 1: Eligible adults who have been treated with ≥ 48 hours of ceftazidime-avibactam in routine practice
  Interventions: Drug: Ceftazidime-avibactam

INTERVENTIONS:
Drug: Ceftazidime-avibactam — Non-Interventional Study

SUMMARY:
The main objective of this non-interventional (retrospective) study is to describe the general treatment patterns, effectiveness, and safety of ceftazidime-avibactam in real-world settings in India. Eligible patients would be adults who have been treated with ≥ 48 hours of ceftazidime-avibactam in routine practice from 01 June 2019 to 01 April 2020. Data of 500 patients will be collected through the abstraction of hospital medical records (electronic) if available or through the individual patient medical record in case electronic records are not available.

ELIGIBILITY:
Inclusion Criteria:

1. more than or equal to 18 years of age
2. Admitted to hospital with documented gram negative infection
3. Has received treatment for atleast 48 hours (complete) with Ceftazidime-Avibactam as a part of his routine clinical management

Exclusion Criteria:

1. The patient is enrolled in any clinical trial of an investigational product
2. Age <18 years
3. Received Ceftazidime avibactam for less than 48 hours.
4. Patient with documented Acinetobacter infection.
5. Patient was a part of named access program or any other interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with documented gram negative infection and treated with Ceftazidime-avibactam for atleast 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- India (8):
  - Fortis Hospital, Bhandup West
  - Apollo Hospital, Chennai
  - Gleneagles Global Hospitals, Chennai
  - Deenanath Mangeshkar Hospital and Research Centre, Erandwane,, PUNE
  - Apollo Hospital, Hyderabad
  - Metro Hospital, Noida
  - Grant Medical Foundation Ruby Hall Clinic, Pune
  - Amri Hospital, WEST Bengal

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=X9001260

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were hospitalized with Gram negative infections and received ceftazidime-avibactam for at least 48 hours in routine clinical practice were included in this retrospective study. Data was collected from electronic health records or participant's medical records. Data was collected for the period from 01-Jun-2019 to 01-Apr-2020 (approximately 10 months).
Groups:
- Ceftazidime-Avibactam: Eligible participants who were hospitalized with Gram negative infections and received ceftazidime-avibactam for at least 48 hours in routine clinical practice were included.
Period: Overall Study
Arm/Group | Ceftazidime-Avibactam
Started | 189
Completed | 189
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants who received ceftazidime-avibactam for at least 48 hours.
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 189
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.6 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 123
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Symptom Improvement at Day 3
Description: The clinical symptom improvement was assessed as per the clinical judgement of the physician and reported as symptom improved and symptom worsened.
Time Frame: Day 3 after ceftazidime-avibactam initiation
Population: Analysis population included all participants who received ceftazidime-avibactam for at least 48 hours. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 103
Participants
  Symptom Improved | 82
  Symptom Worsened | 21

2. Primary Outcome: Number of Participants With Treatment Success at Day 7
Description: The treatment success was defined as resolution of all signs and symptoms of the infection based on the clinician's judgment and the treatment protocol/algorithm followed at the respective centers. The treatment success in terms of clinical outcome was classified as clinical success (resolution of all signs and symptoms of the infection), clinical failure (persistence of signs and symptoms from baseline) and indeterminate (there is not enough information to conclude whether the antibiotic regimen containing ceftazidime-avibactam was a clinical failure or a success).
Time Frame: Day 7 after ceftazidime-avibactam initiation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 83
Participants
  Clinical Success | 66
  Clinical Failure | 12
  Clinical Indeterminate | 5

3. Primary Outcome: Number of Participants With Treatment Success at Day 14 or End of Treatment
Description: as for outcome 2
Time Frame: Day 14 or End of Treatment after ceftazidime-avibactam initiation, whichever was earlier
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 59
Participants
  Clinical Success | 45
  Clinical Failure | 13
  Clinical Indeterminate | 1

4. Primary Outcome: Number of Participants With Microbiological Success at Day 7
Description: Microbiological success was defined as absence of causative pathogen from appropriately obtained specimens at the site of infection (eradication) and repeat cultures were not performed/clinically indicated in a participant who had a clinical response of cure (presumed eradication).
Time Frame: Day 7 after ceftazidime-avibactam initiation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 38
Participants
  Eradication | 31
  Presumed Eradication | 7

5. Primary Outcome: Number of Participants With Microbiological Success at Day 14 or End of Treatment
Description: as for outcome 4
Time Frame: Day 14 or End of Treatment after ceftazidime-avibactam initiation, whichever was earlier
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 41
Participants
  Eradication | 24
  Presumed Eradication | 17

6. Secondary Outcome: Number of Participants Classified According to Source of Infection at Baseline for Which Ceftazidime-Avibactam Was Used
Description: Source of infection included hospital-acquired infection, healthcare-associated infection, and community-acquired infection.
Time Frame: Baseline (before initiation of initial antibiotic therapy)
Population: Analysis population included all participants who received ceftazidime-avibactam for at least 48 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 189
Participants
  Hospital-Acquired Infection | 72
  Healthcare Associated Infection | 65
  Community-Acquired Infection | 52

7. Secondary Outcome: Number of Participants According to Indication at Baseline for Which Ceftazidime-Avibactam Was Used
Description: The indications for use of ceftazidime-avibactam at baseline including urinary tract infection, intra-abdominal infection and nosocomial pneumonia and any other indication were reported.
Time Frame: Baseline (before the initiation of initial antibiotic therapy)
Population: Analysis population included all participants who received ceftazidime-avibactam for at least 48 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 189
Participants
  Urinary Tract Infection | 55
  Intra-abdominal Infection | 30
  Nosocomial Infection | 55
  Others | 49

8. Secondary Outcome: Dose of Ceftazidime - Avibactam
Description: In this outcome measure dose (median of daily dose) of ceftazidime-avibactam was reported till Day 14 or End of treatment whichever was earlier.
Time Frame: Up to Day 14 or End of treatment after ceftazidime-avibactam initiation, whichever was earlier
Population: Analysis population included all participants who received ceftazidime-avibactam for at least 48 hours.
Measure: Median (Full Range); unit: Milligrams
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 189
Milligrams | 2500 [1000 to 2500]

9. Secondary Outcome: Number of Participants According to Frequency of Administration
Description: Number of participants according to frequency of administration (twice daily [BID], once daily [OD] and thrice daily [TID]) of ceftazidime-avibactam is reported in this outcome measure.
Time Frame: Up to Day 14 or End of treatment after ceftazidime-avibactam initiation, whichever was earlier
Population: Analysis population included all participants who received ceftazidime-avibactam for at least 48 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 189
Participants
  BID | 71
  OD | 22
  TID | 96

10. Secondary Outcome: Duration of Administration of Ceftazidime - Avibactam
Time Frame: Up to Day 14 or End of treatment after ceftazidime-avibactam initiation, whichever was earlier
Population: Analysis population included all participants who received ceftazidime-avibactam for at least 48 hours.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 189
Hours | 2.1 (0.8)

11. Secondary Outcome: Total Duration of Therapy of Ceftazidime-Avibactam
Time Frame: Up to Day 14 or End of treatment after ceftazidime-avibactam initiation, whichever was earlier
Population: Analysis population included all participants who received ceftazidime-avibactam for at least 48 hours.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 189
Days | 6.92 (4.1)

12. Secondary Outcome: Number of Participants Who Received Concomitant Antibiotics With Ceftazidime-Avibactam
Time Frame: Up to Day 14 or End of treatment after ceftazidime-avibactam initiation, whichever was earlier
Population: Analysis population included all participants who received ceftazidime-avibactam for at least 48 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 189
Participants | 156

13. Secondary Outcome: Number of Participants With History of Antibiotic Exposure
Time Frame: 90 days prior to current hospital admission
Population: Analysis population included all participants who received ceftazidime-avibactam for at least 48 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 189
Participants | 126

14. Secondary Outcome: Number of Participants According to Identified Gram Negative Organisms
Description: In this outcome measure, the gram-negative organisms identified at baseline was reported. One participant could have more than one gram-negative bacteria identified.
Time Frame: Baseline (before the initiation of initial antibiotic therapy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 84
Participants
  Klebsiella pneumoniae | 57
  Escherichia Coli | 15
  Pseudomonas aeruginosa | 11
  Klebsiella species | 4
  Enterobacter species | 1
  Enterobacter cloacae | 1
  Proteus mirabilis | 1
  Pseudomonas species | 1
  Other | 1

15. Secondary Outcome: Number of Participants With Identified Pathogens Susceptible to Ceftazidime-Avibactam
Time Frame: Baseline (before the initiation of initial antibiotic therapy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 47
Participants | 34

16. Secondary Outcome: Duration of Hospital Stay
Description: Duration of hospital stay was calculated based on 1) total number of consecutive days the participant was treated in the hospital from admission to discharge during their initial hospitalization; 2) the total number of days of hospitalization between diagnosis of infection and discharge; 3) the total number of days the participant was treated in the hospital after ceftazidime-avibactam initiation up to hospital discharge, including the first day of treatment.
Time Frame: Up to 30 days post treatment completion, death or discharge; whichever was first (Up to maximum of 49 days)
Population: Analysis population included all participants who received ceftazidime-avibactam for at least 48 hours.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 189
Days | 23.1 (15.1)

17. Secondary Outcome: Duration of Stay in Intensive Care Unit (ICU)
Description: Intensive care unit length of stay was calculated based on 1) the total number of consecutive or non-consecutive days the participant was treated in the ICU during their initial hospitalization; and 2) the total number of days the participant was treated in the ICU after ceftazidime-avibactam initiation, including the first day of treatment.
Time Frame: Up to 30 days post treatment completion, death or discharge; whichever was first (Up to maximum of 49 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 162
Days | 15.7 (14.3)

18. Secondary Outcome: Number of Participants According to Healthcare Resource Utilization
Description: In this outcome measure number of participants were reported as per their healthcare resource utilization data, abstracted from the participant medical records. Healthcare resources included: mechanical ventilation, computed tomography (CT)/magnetic resonance imaging (MRI), tracheostomy, hemodialysis, surgical intervention, percutaneous procedures and other procedures.
Time Frame: Up to 30 days post treatment completion with ceftazidime-avibactam death or discharge; whichever was first (Up to maximum of 49 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 109
Participants
  Mechanical ventilation | 82
  CT/MRI imaging | 59
  Tracheostomy | 36
  Hemodialysis | 25
  Surgical intervention | 16
  Percutaneous procedures | 5
  Other procedure (Other healthcare resources utilized) | 22

19. Secondary Outcome: Number of Participants With Recurrence of Infection
Description: Number of participants with recurrence of infection during hospital stay, including re-infection and relapse up to 30 days post treatment completion with ceftazidime-avibactam, death or discharge; whichever occurred first was summarized in this outcome measure.
Time Frame: Up to 30 days post treatment completion with ceftazidime-avibactam, death or discharge; whichever was first (Up to maximum of 49 days)
Population: Analysis population included all participants who received ceftazidime-avibactam for at least 48 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 189
Participants | 8

20. Primary Outcome: Number of Participants With Serious Adverse Events and Non-Serious Adverse Events With Explicit Attribution to Ceftazidime-Avibactam
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was any untoward medical occurrence at any dose that: resulted in death, was life threatening (immediate risk of death), required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect. All AEs that did not meet the criteria for "serious" were considered as non-serious. Adverse events with explicit attribution to any Pfizer drug that appeared in the reviewed information (defined per the participant population and study period specified in the protocol) were reported. Explicit attribution was not inferred by temporal relationship between drug administration and an AE, but was based on a causality assessed by a healthcare provider linking drug administration and AE.
Time Frame: as for outcome 19
Population: Analysis population included all participants who received ceftazidime-avibactam for at least 48 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 189
Participants
  Serious adverse events | 0
  Non-serious adverse events | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days post treatment completion with ceftazidime-avibactam, death or discharge; whichever occurred first (up to Day 49)
Arm/Group | Ceftazidime-Avibactam
All-Cause Mortality (participants affected / at risk) | 0/189
Serious Adverse Events (participants affected / at risk) | 0/189
Other Adverse Events (participants affected / at risk) | 0/189

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT04628572/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT04628572/SAP_001.pdf